CLINICAL TRIAL: NCT05531461
Title: COGNITIVE Study- Cognition and Imaging With Tigertriever
Brief Title: Cognition and Imaging With Tigertriever
Acronym: COGNITIVE
Status: Recruiting | Type: Observational
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: COGNITIVE Study
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the COGNITIVE Study is to evaluate whether successful reperfusion with Tigertriever is associated with cognitive benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with large vessel occlusion (LVO) and treated with the Tigertriever, as indicated per the approved IFU.
2. Tigertriever was used as the first line treatment in the target vessel.
3. A signed informed consent.
4. Age 18-75 years (inclusive).
5. No known significant pre-stroke disability (pre-stroke mRS 0 or 1).

Exclusion Criteria:

1. Use of any other IA recanalization device prior to the Tigertriever in the target vessel, including aspiration catheter.
2. Evidence of acute brain hemorrhage on CT and/or MRI at admission.
3. Prior hemorrhage, stroke, thrombolysis, and/or endovascular therapy in the last 3 months.
4. Probable cerebral amyloid angiopathy.
5. Pre-stroke diagnosed dementia and/or prescribed cholinesterase inhibitors.
6. Pre-stroke diagnosed and/or currently treated major depression.
7. Pre-stroke learning or intellectual disability.
8. Anticipated inability to obtain 6-month follow-up assessments.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The COGNITIVE Study will include male or female subjects age 18-75 who present with LVO and treated with the Tigertriever as indicated per approved IFU.
Sampling Method: Probability Sample
Enrollment: 424 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Association between successful reperfusion* and cognitive benefit** | 180 days post treatment
  *successful reperfusion is defined as eTICI ≥2b50 with the Tigertriever device.
  * Cognitive benefit is defined as change in Montreal Cognitive Assessment (MoCA) of 1.5 Standard Deviations (SD) from 4 days post treatment (or discharge if earlier) and 180 days post treatment; or MoCA ≥26 at 180 days post treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Los Angeles, California
  - Corewell Health Research Institute, Grand Rapids, Michigan
  - Westchester Medical Center, New York, New York